CLINICAL TRIAL: NCT00056524
Title: An Open-Label Multicenter Study to Assess the Safety of AVP-923 in the Treatment of Patients With Pseudobulbar Affect.
Brief Title: Safety Study of AVP-923 in the Treatment of IEED (Involuntary Emotional Expression Disorder) Also Known as Pseudobulbar Affect (Episodes of Uncontrolled Crying and/or Laughter)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-AVR-107; AVP-923
Record Dates: First submitted 2003-03-15; First posted 2003-03-18 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Alzheimer's Disease; Stroke; Parkinson's Disease; Traumatic Brain Injury
Keywords: ALS; MS; CNS; AD; TBI; Dextromethorphan; IEED; Emotional
MeSH Terms: conditions — Alzheimer Disease; Stroke; Parkinson Disease; Brain Injuries, Traumatic | interventions — dextromethorphan - quinidine combination

INTERVENTIONS:
Drug: AVP-923

SUMMARY:
The purpose of this study is to evaluate the long-term safety of AVP-923 in the treatment of Involuntary Emotional Expression Disorder (IEED) also known as Pseudobulbar Affect (episodes of uncontrolled crying and/or laughter).

DETAILED DESCRIPTION:
This is an "open label" study which means there is no placebo group. Each subject enrolled into the study will receive AVP-923.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age, inclusive
* Clinical diagnosis of PBA (pseudobulbar affect)
* If female, must not be pregnant or breast feeding

Exclusion Criteria:

* Sensitivity to quinidine or any opiate drugs
* Current or prior history of major psychiatric disturbance
* Currently participated in a trial within the past 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2003-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
emotional control

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Center for Neurologic Study, La Jolla, California
  - UCLA School of Medicine, Los Angeles, California
  - UCSF, San Francisco, California
  - Research Center for Clinical Studies, Inc., Darien, Connecticut
  - George Washington University Medical Faculty Assoc., Washington D.C., District of Columbia
  - Neurological Associates, Fort Lauderdale, Florida
  - University of Miami Dept. of Neurology, Miami, Florida
  - Miami Jewish Home & Hospital for the Aged, Miami, Florida
  - Allied Clinical Trials, Miami, Florida
  - Renstar Medical Research, Plantation, Florida
  - Suncoast Neuroscience Associates Inc., St. Petersburg, Florida
  - Tampa, Florida
  - Neurology & Headache Specialist of Atlanta, L.L.C., Decatur, Georgia
  - Consultants in Neurology LTD, Northbrook, Illinois
  - Advanced Neurology Specialists, Great Falls, Montana
  - Neurological Associates, P.C., Lincoln, Nebraska
  - Upstate Clinical Research, Albany, New York
  - DENT Neurologic Group L.L.P., Amherst, New York
  - Hospital for Joint Diseases MS Care Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Raleigh Neurology Associates, PA, Raleigh, North Carolina
  - NeuroCare Center, Inc., Canton, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University Memory and Aging Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Clinical Pharmaceutical Trials, Inc., Tulsa, Oklahoma
  - Lehigh Valley Neurosciences and Pain Research Center, Allentown, Pennsylvania
  - Westmoreland Neurology, Greensburg, Pennsylvania
  - Jenkintown, Pennsylvania
  - MCP-Hahnemann University, Philadelphia, Pennsylvania
  - Penn Neurological Institute, Philadelphia, Pennsylvania
  - Neurological Associates of Delaware Valley, Upland, Pennsylvania
  - Claghorn-Lesem Research Clinic, Bellaire, Texas
  - Methodist Neurological Institute, Houston, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Neurology and Neurosurgery Associates of Tacoma, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Pattee GL, Wymer JP, Lomen-Hoerth C, Appel SH, Formella AE, Pope LE. An open-label multicenter study to assess the safety of dextromethorphan/quinidine in patients with pseudobulbar affect associated with a range of underlying neurological conditions. Curr Med Res Opin. 2014 Nov;30(11):2255-65. doi: 10.1185/03007995.2014.940040. Epub 2014 Jul 28. PMID 25062507